CLINICAL TRIAL: NCT06798298
Title: A Long-Term Follow-up Protocol for Participants Treated With Gene Modified T Cells
Brief Title: A Safety and Efficacy Long-Term Follow-up Study of Adult Participants Treated With Gene Modified T Cells
Status: Recruiting | Type: Observational
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: LTF-01
Record Dates: First submitted 2025-01-09; First posted 2025-01-29 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Long Term Safety Following GM T Cell Therapy
Keywords: GM T cell therapy; Replication Competent Lentivirus (RCL)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- GM T cell population: Participants exposed to gene modified T cell therapy on a 2seventy bio (prior to April 2024) or Regeneron Pharmaceuticals sponsored study
  Interventions: Genetic: Non-interventional

INTERVENTIONS:
Genetic: Non-interventional — No study drug administered. Long-term follow-up only.

SUMMARY:
This is a prospective study for the Long-Term Follow-Up (LTFU) of safety and efficacy of all participants exposed to gene modified (GM) T cell therapy in accordance with Health Authorities' guidance for participants treated with gene therapy products.

Participants who received at least one infusion of gene modified T cells in a 2seventy bio (prior to April 2024) or Regeneron Pharmaceuticals sponsored study will be asked to participate in this LTFU protocol, upon either premature discontinuation from, or completion of the parent treatment protocol.

Participants enrolled in this LTFU protocol will have safety assessments, laboratory evaluations, and complete patient-reported outcome (PRO) questionnaires at scheduled intervals as applicable.

ELIGIBILITY:
Inclusion Criteria:

1. All participants who received at least one GM T cell infusion in a previous 2seventy bio (prior to April 2024) or Regeneron Pharmaceuticals sponsored study, and have completed the post-treatment follow-up period on the parent treatment protocol, or discontinued follow-up on the parent protocol after completing at least 6 months of safety monitoring, as applicable.
2. Participant (and legal representative, when applicable) must understand and voluntarily sign an Informed Consent Form (ICF)/Informed Assent Form (IAF) prior to any study related assessments/procedures being conducted.

Exclusion Criteria:

Not applicable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Enrolled participants will be determined by the number of participants participating in GM T cell 2seventy bio (prior to April 2024) and Regeneron Pharmaceuticals sponsored studies consenting to participate in the LTFU study.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-11-10 (Actual); Primary Completion 2040-06-17 (Estimated); Study Completion 2040-06-17 (Estimated)

PRIMARY OUTCOMES:
Incidence of delayed adverse events considered at least possibly related to prior gene modified T cell therapy | Up to 15 years
Persistence of gene modified T cells | Up to 15 years
Analysis of vector integration sites | Up to 15 years
Incidence of RCL | Up to 15 years
Disease progression status | Up to 15 years
  To assess long-term efficacy following treatment with gene modified T cells
Date of disease progression | Up to 15 years
Survival status | Up to 15 years

SECONDARY OUTCOMES:
Health-Related Quality of Life (HRQoL) Changes | Up to 5 years
  Assessed using instruments administered in the parent treatment protocol

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (1):
- Tennessee Oncology, Nashville, Tennessee, United States